CLINICAL TRIAL: NCT05992805
Title: ScanNav Anatomy PNB Data Collection Study
Status: Completed | Type: Observational
Sponsor: IntelligentUltrasound Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: IU2023_AG_11
Record Dates: First submitted 2023-03-27; First posted 2023-08-15 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Volunteer Participants: Volunteer participants being scanned by a qualified clinician using various ultrasound machines.
  Interventions: Other: N/A - non-interventional study

INTERVENTIONS:
Other: N/A - non-interventional study — N/A - non-interventional study. Data collection only.

SUMMARY:
Study to gather additional data for AI-driven medical device, ScanNav Anatomy PNB.

DETAILED DESCRIPTION:
Volunteer study to gather additional ultrasound training and/or validation data for Artificial Intelligence (AI)-algorithms used in the medical device ScanNav Anatomy PNB.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age;
2. Able to comprehend and sign the Informed Consent prior to enrolment in the study.

Exclusion Criteria:

1. Aged <18 years of age;
2. Unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Training and/or validation data (in the form of recorded ultrasound scans) | 6 months
  Ultrasound scans to be used for training and/or validation of AI models developed in-house to assist ultrasound-guided regional anaesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Hodge House, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No